CLINICAL TRIAL: NCT04226664
Title: Bariatric Surgery for the Reduction of cArdioVascular Events Feasibility Randomized Controlled Trial (BRAVE)
Brief Title: Bariatric Surgery for the Reduction of cArdioVascular Events Feasibility Trial
Acronym: BRAVE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Population Health Research Institute (Other); St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 8047
Record Dates: First submitted 2020-01-03; First posted 2020-01-13 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Obesity, Morbid; Cardiovascular Diseases
Keywords: Bariatric Surgery
MeSH Terms: conditions — Obesity, Morbid; Cardiovascular Diseases | interventions — Bariatric Surgery

STUDY DESIGN:
Intervention Model Description: Individuals who meet study eligibility criteria will be randomized in 1:1 fashion to bariatric surgery (intervention arm) or MWM (control arm).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): Bariatric surgery will consist of laparoscopic Roux-en-Y gastric bypass or sleeve gastrectomy performed at the discretion of the surgeon and according to local standards.
  Interventions: Procedure: Bariatric surgery
- Control (No Intervention): Medical Weight Management (MWM) corresponds to the standard medical practice for weight loss that is available at the local participating centre, and thus reflects the local standard of care.

INTERVENTIONS:
Procedure: Bariatric surgery — Although there may be slight variation by centre, Gastric Bypass generally involves creation of a 30-50 cc stomach pouch, which is anastamosed with a Roux limb of jejunum 75-100 cm in length and a biliary limb of 20-30 cm in length. The operation creates a small gastric pouch, with nutrients bypassing the duodenum and proximal jejunum. Sleeve Gastrectomy involves decreasing the size of the stomach to approximately 15% of its original size by resecting a large portion of the stomach along the greater curvature.
  Arms: Intervention

SUMMARY:
Pilot multicentre, open-label, parallel-arm randomized controlled trial (RCT) of 60 patients to demonstrate the feasibility of enrolling patients with high-risk cardiovascular disease (CVD) into an RCT of bariatric surgery versus medical weight management (MWM).

DETAILED DESCRIPTION:
STUDY OBJECTIVE The primary objective of this pilot study is to assess the feasibility of an RCT of bariatric surgery compared to MWM in patients with morbid obesity and high-risk CVD. If we can demonstrate that this trial is feasible, the next step would be to conduct a large-scale RCT to evaluate the efficacy of bariatric surgery for the reduction of cardiovascular complications in this patient population.

STUDY AIMS:

1. To demonstrate that enrolment of high-risk CVD patients into a bariatric surgery RCT is feasible.
2. To show that it is feasible to perform bariatric surgery in >80% of patients in the intervention arm within 30 days of randomization.
3. To obtain preliminary information on the perioperative risks of bariatric surgery in patients with high-risk CVD.

STUDY HYPOTHESES Study enrollment will be feasible at a rate of at least 1.25 patients per centre per month. Timely delivery of the intervention is possible, with >80% of patients undergoing bariatric surgery within 30 days of randomization. The rate of crossover between the control and intervention arms will be low at <2.5% per year. 30-day mortality rates in the intervention group will be comparable to that of an age and gender matched cohort without CVD who had bariatric surgery at the 2 study sites during the study period.

DESIGN The present study is a multicentre, open-label, parallel-arm feasibility RCT with blinded endpoint assessment (PROBE design) of bariatric surgery compared to MWM in patients with morbid obesity and high-risk CVD.

Individuals who meet study eligibility criteria will be randomized in 1:1 fashion to bariatric surgery (intervention arm) or MWM (control arm). Bariatric surgery will consist of laparoscopic Roux-en-Y gastric bypass or sleeve gastrectomy, performed at the discretion of the surgeon and according to local standards.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index >35 kg/m2
2. Age ≥18 years
3. High-risk CVD, defined as the presence of any one of the following:

   1. History of MI, multi-vessel percutaneous coronary intervention or multi-vessel coronary artery bypass grafting; OR
   2. Coronary artery disease (CAD) with documented stenoses ≥50% in 2 or more major coronary arteries; OR
   3. Symptomatic HF (New York Heart Association class ≥2) on optimal HF therapy for ≥3 months, AND documented HF hospitalization within the last 12 months, OR baseline N-terminal pro B-type natriuretic peptide (NT-pro BNP) >400 pg/ml;44, 45 OR
   4. Documented AF with CHA2DS2-VASc stroke risk score (congestive heart failure/ left ventricular dysfunction, hypertension, age ≥ 75 years [2 points], diabetes, history of stroke/ transient ischemic attack [2 points], vascular disease, age 65-74 years and female sex) of ≥2; OR
   5. History of ischemic stroke; OR
   6. Peripheral artery disease, defined as prior aorto-femoral bypass surgery, limb bypass surgery, or percutaneous transluminal angioplasty revascularization of the iliac, infra-inguinal arteries or carotids; or limb or foot amputation for arterial vascular disease; or ≥50% carotid or peripheral artery stenosis
4. Patient is deemed eligible to undergo bariatric surgery according to local practice guidelines

Exclusion Criteria:

1. Hospital admission for HF within 30 days of enrolment
2. Myocardial infarction, stroke or coronary revascularization in prior 30 days.
3. Percutaneous coronary intervention with a drug eluting stent in prior 90 days.
4. Pregnancy
5. Contraindication to bariatric surgery (atrophic gastritis, diabetes mellitus type 1, prior laparotomy, liver cirrhosis with portal hypertension, uncontrolled drug or alcohol dependence, prior bariatric surgery, massive ventral hernia, severe chronic obstructive pulmonary disease)
6. Life expectancy <2 years from non-cardiovascular causes.
7. Risk of general anesthesia deemed too excessive
8. Current drug or alcohol dependency (within 6 months of referral)
9. Recent major cancer (life threatening, within last 2 years)
10. Untreated or inadequately treated psychiatric illness
11. Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-30 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Recruitment rate | 24 months (or when recruitment is complete)
  Recruitment rate (target of 60 patients over 24 months or 1.25 patients per centre per month)
Time to intervention administration | 30 days
  Target of bariatric surgery performed within 30 days of randomization in >80%
Crossover rate | At study completion (an average of 1.5 years follow-up)
  Crossover rate between control and intervention arm

SECONDARY OUTCOMES:
Change in weight at 1 year | 12 months
  Change in weight in kilograms at 1 year
Change in BMI at 1 year | 12 months
  BMI (kg/m^2) will be calculated using weight in kg at 1 year, and height
Composite outcome of cardiovascular mortality, myocardial infarction (MI), stroke and hospitalization for heart failure (HF) | 12 months, and through study completion (an average of 1.5 years follow-up)
  Composite outcome of cardiovascular mortality, myocardial infarction, stroke and hospitalization for heart failure
Change in percent excess weight loss (%) at 1 year | 12 months
  Excess weight loss is a standard outcome measure in obesity research. It is calculated as the percentage of excess body weight lost after surgery. Excess body weight (kg) is calculated as current weight (kg) minus ideal body weight (kg) for a given height. Ideal body weight (kg) is taken from standardized tables.
Change in New York Heart Association (NYHA) Functional Classification at 1 year | 12 months
  NYHA Class is a standardized classification system for severity of heart failure symptoms, and ranges from class I to class IV, with IV being the most severe symptoms and class.
Change in 6-minute walk test distance (m) at 1 year | 12 months
  The 6 Minute Walk Test is an exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome. Longer distances indicate better performance.
Change in 36-Item Short Form Survey (SF-36) questionnaire score at 1 year | 12 months
  The SF-36 is a measure of health-related quality-of-life. It includes eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state.
Change in EuroQuol (EQ-5D-5L) quality of life questionnaire score at 1 year | 12 months
  EQ-5D-5L is a standardized instrument for measuring health status, which includes a descriptive system asking about 5 health dimensions as well as an evaluation of overall health status with a visual analogue scale. The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels from which respondents choose one response: no problems, slight problems, moderate problems, severe problems and extreme problems. The visual analogue scale asks individuals to mark their health status on the day of the interview on a 20 cm vertical scale with end points of 0 and 100. Zero corresponds to " the worst health you can imagine", and 100 corresponds to "the best health you can imagine".
Number of participants with new onset Atrial Fibrillation (AF) at 1 year | 12 months, and through study completion (an average of 1.5 years follow-up)
  Will determine the number of participants who receive a new clinical diagnosis of AF during the study follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Wong, MD MPH FRCPC, Principal Investigator — PHRI, Hamilton Health Sciences, McMaster University; Aristithes Doumouras, MD MPH FRCSC, Principal Investigator — St. Joseph's Healthcare, McMaster University
Locations (1):
- St. Joseph's Healthcare Hamilton, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Population Health Research Institute — http://www.phri.ca/
- See also: St. Joseph's Heathcare Hamilton Bariatric Surgery Program — https://www.stjoes.ca/hospital-services/surgical-services/bariatric-surgery